CLINICAL TRIAL: NCT01491672
Title: An Open-label, Multicenter Phase II Study to Examine the Efficacy and Safety of Everolimus as Second-line Therapy in the Treatment of Patients With Metastatic Renal Cell Carcinoma
Brief Title: Everolimus as Second-line Therapy in Metastatic Renal Cell Carcinoma
Acronym: RECORD-4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001L2404; 2010-020447-13 (EudraCT Number)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma; Second Line; Everolimus; RAD001
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): Participants, received RAD001 10 mg orally once daily.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Study drug was supplied as 5 mg tablets in blister packs.
  Other Names: Everolimus

SUMMARY:
This study will evaluate everolimus as second-line therapy in patients with metastatic renal cell carcinoma. Each patient will be enrolled and stratified in one of three cohorts based upon their first-line therapy: 1) prior cytokines, 2) prior sunitinib, or 3) prior anti-VEGF therapy other than sunitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Patients with advanced renal cell carcinoma of a histological or cytological confirmation of clear cell (or with a component of clear cell) renal carcinoma that have previously progressed on or were intolerant to first-line therapy with sunitinib, sorafenib, pazopanib, axitinib, bevacizumab, or cytokine therapy.
3. Patients must have had prior nephrectomy (partial or total).
4. Patients with at least one measurable lesion at baseline as per the RECIST 1.0 criteria. If skin lesions are reported as target lesions, they should be documented (at baseline and at every physical exam) using color photography and a measuring device (such as a caliper) in clear focus to allow the size of the lesion(s) to be determined from the photograph.
5. Patients with a Karnofsky Performance Status ≥ 70%.
6. Adequate bone marrow function as shown by:

   1. ANC ≥ 1.5 x 109/L,
   2. Platelets ≥ 100 x 109/L,
   3. Hemoglobin >9 g/dL
7. Adequate liver function as shown by:

   1. Serum bilirubin ≤ 1.5 x ULN,
   2. ALT and AST ≤ 2.5 x ULN. Patients with known liver metastases may enroll if their AST and ALT ≤ 5 x ULN,
   3. INR < 1.3 (INR < 3 in patients treated with anticoagulants)
8. Adequate renal function: serum creatinine ≤ 2.0 x ULN.
9. Fasting serum cholesterol ≤300 mg/dl OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5 x ULN.
10. Written informed consent obtained before any trial related activity and according to local guidelines.

Exclusion Criteria:

1. Patients with brain metastases.
2. Patients within 4 weeks post-major surgery (e.g., intra-thoracic, intra-abdominal or intrapelvic), open biopsy, or significant traumatic injury to avoid wound healing complications.

   Minor procedures and percutaneous biopsies or placement of vascular access device require 7 days prior to study entry.
3. Patients in anticipation of the need for major surgical procedure during the course of the study.
4. Patients who had radiation therapy within 4 weeks prior to start of study treatment (palliative radiotherapy to bone lesions allowed up to 2 weeks prior to study treatment start).
5. Patients with a serious non-healing wound, ulcer, or bone fracture.
6. Patients with a history of seizure(s) not controlled with standard medical therapy.
7. Patients who have received more than one prior treatment regimen for metastatic renalcell carcinoma
8. Patients who have received adjuvant therapy for RCC
9. Patients who have previously received systemic mTOR inhibitors (eg, sirolimus, temsirolimus, everolimus)
10. Patients with a known hypersensitivity to everolimus or other rapamycins (eg, sirolimus, temsirolimus) or to its excipients.
11. History or clinical evidence of central nervous system (CNS) metastases.
12. Clinically significant gastrointestinal abnormalities including, but not limited to:

    1. Malabsorption syndrome:
    2. Major resection of the stomach or small bowel that could affect the absorption of study drug
    3. Active peptic ulcer disease
    4. Inflammatory bowel disease:

    i. Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation ii. History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
13. Patients with a known history of HIV seropositivity. Screening for HIV infection at baseline is not required.
14. Active bleeding diathesis
15. Uncontrolled diabetes mellitus as defined by fasting serum glucose > 2.0 x ULN.
16. Patients who have any severe and/or uncontrolled medical conditions such as:

    1. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction

       ≤ 6 months prior to enrollment, serious uncontrolled cardiac arrhythmia,
    2. active or uncontrolled severe infection,
    3. history of invasive fungal infections,
    4. severe hepatic impairment (Child-Pugh class C),
    5. severely impaired lung function
17. History of cerebrovascular accident (CVA) including transient ischemic attack (TIA) ≤ 6 months before start of study treatment.
18. History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
19. Patients who have a history of another primary malignancy and off treatment for ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix or breast, and localized cancer of the bladder (T1) and prostate (T1 - T2).
20. Female patients who are pregnant or nursing (lactating).
21. Adults of reproductive potential who are not using effective birth control methods.

    Adequate contraceptives must be used throughout the trial and for 8 weeks after last study drug administration in female patients. Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to first administration of study drug.
22. Patients who are using other investigational agents or who had received investigational drugs ≤ 2 weeks prior to study treatment start. This should not include sunitinib, sorafenib, axitinib, pazopanib and cytokines.
23. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Argentina (2):
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Rio Negro, Viedma
- Brazil (3):
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sofia, Bulgaria
- China (5):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Russia (4):
  - Novartis Investigative Site, Leningrad Region, Russia
  - Novartis Investigative Site, Moscow, Russia
  - Novartis Investigative Site, Nizhny Novgorod, Russia
  - Novartis Investigative Site, Obninsk, Russia

REFERENCES:
- [Derived] Yang L, Alyasova A, Ye D, Ridolfi A, Dezzani L, Motzer RJ. RECORD-4 multicenter phase 2 trial of second-line everolimus in patients with metastatic renal cell carcinoma: Asian versus non-Asian population subanalysis. BMC Cancer. 2018 Feb 17;18(1):195. doi: 10.1186/s12885-018-4091-5. PMID 29454306
- [Derived] Motzer RJ, Alyasova A, Ye D, Karpenko A, Li H, Alekseev B, Xie L, Kurteva G, Kowalyszyn R, Karyakin O, Neron Y, Cosgriff T, Collins L, Brechenmacher T, Lin C, Morgan L, Yang L. Phase II trial of second-line everolimus in patients with metastatic renal cell carcinoma (RECORD-4). Ann Oncol. 2016 Mar;27(3):441-8. doi: 10.1093/annonc/mdv612. Epub 2015 Dec 17. PMID 26681676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study where all eligible participants were enrolled into one of 3 cohorts based upon prior first-line therapy.
Groups:
- Prior Sunitinib: Participants, who received prior sunitinib therapy, received RAD001 10 mg orally once daily.
- Other Prior Vascular Endothelial Growth Factor (VEGF): Participants, who received prior anti-VEGF other than sunitinib, received RAD001 10 mg orally once daily.
- Prior Cytokines: Participants, who received prior cytokine therapy, received RAD001 10 mg orally once daily.
Period: Overall Study
Arm/Group | Prior Sunitinib | Other Prior Vascular Endothelial Growth Factor (VEGF) | Prior Cytokines
Started | 58 | 62 (1 participant died prior to treatment initiation.) | 14
Safety Set | 58 | 61 | 14
Completed | 2 | 2 | 3
Not Completed | 56 | 60 | 11
Not completed — Lost to Follow-up | 0 | 4 | 1
Not completed — Withdrawal by Subject | 6 | 7 | 0
Not completed — Adverse Event | 8 | 10 | 4
Not completed — Disease progression | 42 | 34 | 6
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Death | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior Sunitinib | Other Prior Vascular Endothelial Growth Factor (VEGF) | Prior Cytokines | Total
Number analyzed (Participants) | 58 | 62 | 14 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (12.06) | 56.5 (11.14) | 60.3 (10.59) | 56.7 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 6 | 43
  Male | 43 | 40 | 8 | 91

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) - All Participants
Description: PFS during second-line treatment was defined as the time from the date of enrollment to the date of the first documented disease progression or death due to any cause. The primary analysis of PFS was based on a local radiology review of CT scans and MRI collected until the participant experienced disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.0.
Time Frame: 20 months
Population: The full analysis set (FAS) was used. It included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Participants: All participants received RAD001 10 mg daily.
Arm/Group | All Participants
Number analyzed (Participants) | 134
months | 7.4 [5.6 to 10.5]

2. Secondary Outcome: Duration of PFS for Each First-line Treatment Cohort
Description: Duration of PFS during second-line treatment was defined as the time from the date of enrollment to the date of the first documented disease progression or death due to any cause. Participants' assessment was based on the local radiological data according to the RECIST 1.0 Criteria.
Time Frame: 20 months
Population: The FAS was used. It included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prior Sunitinib | Other Prior Vascular Endothelial Growth Factor (VEGF) | Prior Cytokines
Number analyzed (Participants) | 58 | 62 | 14
months | 5.6 [3.7 to 11.3] | 7.8 [5.7 to 11.0] | 12.9 [2.6 to NA] — The upper limit was not estimable using the Kaplan Meier (KM) method as a result of too few events.

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of enrollment to date of death due to any cause.
Time Frame: 28 months
Population: The FAS was used. It included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prior Sunitinib | Other Prior Vascular Endothelial Growth Factor (VEGF) | Prior Cytokines | All Participants
Number analyzed (Participants) | 58 | 62 | 14 | 134
months | 23.8 [13.7 to NA] — The upper limit was not estimable using the Kaplan Meier (KM) method as a result of too few events. | 17.2 [11.9 to NA] — The upper limit was not estimable using the Kaplan Meier (KM) method as a result of too few events. | NA [15.9 to NA] — The upper limit was not estimable using the Kaplan Meier (KM) method as a result of too few events. | 23.8 [17.0 to NA] — The upper limit was not estimable using the Kaplan Meier (KM) method as a result of too few events.

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) or stable disease based on the local radiological data according to the RECIST 1.0 criteria.
Time Frame: 20 months
Population: The FAS was used. It included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Prior Sunitinib | Other Prior Vascular Endothelial Growth Factor (VEGF) | Prior Cytokines | All Participants
Number analyzed (Participants) | 58 | 62 | 14 | 134
Participants | 41 | 48 | 11 | 100

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants with best overall response of CR or PR based on the local radiological data according to the RECIST 1.0 Criteria
Time Frame: 20 months
Population: The FAS was used. It included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Prior Sunitinib | Other Prior Vascular Endothelial Growth Factor (VEGF) | Prior Cytokines | All Participants
Number analyzed (Participants) | 58 | 62 | 14 | 134
Participants | 4 | 3 | 3 | 10

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from the first occurrence of PR or CR (as per local radiological review) until the date of the first documented disease progression or death due to underlying cancer.
Time Frame: 20 months
Population: The FAS was considered for this analysis. The FAS included all enrolled participants. Only participants who achieved a CR or PR were analyzed. Therefore, actual n=4,3,3,10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prior Sunitinib | Other Prior Vascular Endothelial Growth Factor (VEGF) | Prior Cytokines | All Participants
Number analyzed (Participants) | 58 | 62 | 14 | 134
months | 10.8 [9.2 to NA] — The upper limit was not estimable using the Kaplan Meier (KM) method as a result of too few events. | 7.4 [3.3 to 9.2] | 9.2 [NA to NA] — The lower and upper limits were not estimable using the Kaplan Meier (KM) method as a result of too few events. | 9.2 [3.3 to NA] — The upper limit was not estimable using the Kaplan Meier (KM) method as a result of too few events.

ADVERSE EVENTS:
Groups:
- Other Prior Anti VEGF: Participants, who received prior anti-VEGF other than sunitinib, received RAD001 10 mg orally once daily.
Arm/Group | Prior Sunitinib | Other Prior Anti VEGF | Prior Cytokines
Serious Adverse Events (participants affected / at risk) | 13/58 | 16/61 | 3/14
Other Adverse Events (participants affected / at risk) | 28/58 | 33/61 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Sunitinib (N=58) | Other Prior Anti VEGF (N=61) | Prior Cytokines (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 2 | 0
Sudden death (General disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
X-ray with contrast upper gastrointestinal tract abnormal (Investigations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Sunitinib (N=58) | Other Prior Anti VEGF (N=61) | Prior Cytokines (N=14)
Anaemia (Blood and lymphatic system disorders) | 8 | 8 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 8 | 5
Fatigue (General disorders) | 0 | 2 | 1
General physical health deterioration (General disorders) | 3 | 1 | 0
Pyrexia (General disorders) | 2 | 5 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 1
Blood pressure increased (Investigations) | 0 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 1
Hepatitis B DNA increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 4 | 2
Proteinuria (Renal and urinary disorders) | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.